CLINICAL TRIAL: NCT00684892
Title: A Safety and Feasibility Study of the Chartis System in Subjects With Heterogeneous Emphysema Prior to Endobronchial Lung Volume Reduction (ELVR)
Brief Title: Safety and Feasibility Study of the Chartis System With Heterogeneous Emphysema Prior to Endobronchial Lung Volume Reduction (ELVR)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Pulmonx Corporation (Industry)
Responsible Party: Carol Anne Yarbrough, RN, Director, Clinical Affairs, Pulmonx, Inc.
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PRT01029
Record Dates: First submitted 2008-05-23; First posted 2008-05-28 (Estimated); Last update posted 2009-01-22 (Estimated); Status verified 2009-01

CONDITIONS: Heterogeneous Emphysema
Keywords: Emphysema; Endobronchial Lung Volume Reduction
MeSH Terms: conditions — Emphysema

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Device: Chartis System

INTERVENTIONS:
Device: Chartis System — Assessment of airway flow and pressure

SUMMARY:
The purpose of this study is to evaluate the safety and feasibility of the Chartis System in measuring air flow and pressures in isolated lung compartments in emphysema patients prior to endobronchial lung volume reduction (ELVR).

ELIGIBILITY:
Inclusion Criteria:

* Heterogeneous emphysema as determined by high-resolution CT scan
* Scheduled for clinically indicated ELVR procedure

Exclusion Criteria:

* Hyperexcretive chronic bronchitis or excessive sputum secretion
* Active pulmonary infection
* Active asthma or lung hyper-responsiveness

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2008-05; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
Adverse events | Until end of study procedure

SECONDARY OUTCOMES:
Technical success | During procedure and up 1 week post procedure

CONTACTS AND LOCATIONS:
Overall Officials: Felix Herth, MD, Principal Investigator — Thoraxklinik am Universitatsklinikum Heidelberg
Locations (1):
- Thoraxklinik am Universitatsklinikum Heidelberg, Heidelberg, Germany